CLINICAL TRIAL: NCT03883581
Title: Impact of Nuedexta on Bulbar Physiology and Function in ALS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Holy Cross Hospital, Florida (Other); ALS Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201802938; OCR20392 (Other: UF OnCore)
Record Dates: First submitted 2019-03-12; First posted 2019-03-21 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: bulbar dysfunction
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Dextromethorphan; Quinidine; dextromethorphan - quinidine combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ALS individuals with bulbar dysfunction (Experimental): Participants enrolled in this group will be prescribed dextromethorphan HBr and quinidine sulfate (Nuedexta) as recommended by their treating neurologist. 20 mg dextromethorphan HBr and 10mg quinidine sulfate will be administered orally with 1 capsule every day for the initial 7 days followed by 1 capsule every 12 hours for the remaining 23 days of the study. Participants will be evaluated 30 days apart to determine the impact of treatment.
  Interventions: Drug: dextromethorphan HBr and quinidine sulfate

INTERVENTIONS:
Drug: dextromethorphan HBr and quinidine sulfate — All eligible and enrolled study participants will be administered the study drug, Nuedexta, as recommended by their treating neurologists.The drug will be administered per the efficacy and safety protocol, with no changes in administration method or recommended dose for individuals with ALS. Prior to commencing treatment with Nuedexta, participants will undergo a comprehensive bulbar evaluation of swallowing, airway protection, speech functions, and complete validated patient-reported surveys. Following 30 days of Nuedexta treatment, participants will be e-evaluated using the same battery of assessments.
  Other Names: Nuedexta

SUMMARY:
Nuedexta is FDA approved for the treatment of pseudobulbar affect in ALS patients and anecdotal reports of improvements in speech, salivation or swallowing have been reported. However, no prospective study has been conducted to comprehensively examine and determine the physiologic impact of Nuedexta on both speech and swallowing physiology in a large group of ALS individuals. These data are needed in order to provide evidence-based guidance to the management of bulbar dysfunction in ALS.

DETAILED DESCRIPTION:
Although advances in the management of bulbar dysfunction in ALS have been disappointing, recent interest has surfaced regarding the therapeutic potential of a pharmaceutical agent, Nuedexta (dextromethorphan HBr and quinidine sulfate), for the treatment of bulbar symptomology in individuals with ALS. Although Nuedexta received approval from the Food and Drug Administration (FDA) to target symptoms of pseudobulbar affect (PBA) in ALS; anecdotal reports of improvements in speech, salivation or swallowing were reported from Neurologists treating ALS individuals who were administered Nuedexta. Subsequently, a Phase II clinical trial was conducted that reported improvements in speech, swallowing and salivation following 30-days of Nuedexta treatment. One serious limitation of this study, however, is the fact that the primary outcome employed was a perceptual patient-report scale (PRO) (Center for Neurological Study Bulbar Function Scale, CNS-BFS), with no objective physiologic outcomes to confirm actual change in bulbar physiology. The absence of any objective clinical physiologic outcomes is particularly important when examining effects of Nuedexta, given that it contains selective serotonin reuptake inhibitors (SSRIs), or serotonergic antidepressants, that can impact the regulation of emotional expression, feelings of wellbeing and modulation of depression (all known to impact the response an individual will provide on a PRO measure). Furthermore, findings based on PRO's must be validated with studies that utilize objective physiologic outcomes of speech and swallowing function. Great excitement exists regarding the potential impact of Nuedexta on bulbar function in ALS with many neurologists prescribing Nuedexta to treat these symptoms in ALS patients. To date, however; no data exists to examine and determine the physiologic impact of Nuedexta on speech or swallowing physiology. These data are needed in order to validate the initial patient-reported outcomes of the Phase II clinical trial and to provide evidence-based guidance to the management of bulbar dysfunction in ALS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable-definite ALS (El-Escorial Criterion);
* ALSFRS-R Bulbar subscale score <10
* Bamboo oral reading speaking rate <140 words per minute
* No allergies to barium sulfate.

Exclusion Criteria:

* Treatment for sialorrhea within the past 3 months that includes either Botox or radiation treatment
* Participation in another disease modifying study targeting bulbar or cough function
* Use of invasive mechanical ventilation/presence of tracheostomy
* Advanced frontotemporal dementia or significant cognitive dysfunction
* Nil per oral status for feeding (i.e., NPO, nothing by mouth)
* Previously prescribed Nuedexta. Additionally, if participants are taking Riluzole or other medications to control sialorrhea, they must be on a stable dose for at least 30 days prior to enrollment in the current study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Tabor, PhD, Principal Investigator — Phil Smith Neuroscience Institute at Holy Cross Hospital; Emily Plowman, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Phil Smith Neuroscience Institute at Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment and enrollment took place at the Phil Smith Neuroscience Institute. Recruitment began in July 25, 2019 and ended in August 2021
Period: Overall Study
Arm/Group | ALS Individuals With Bulbar Dysfunction
Started | 28
Completed | 24
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | ALS Individuals With Bulbar Dysfunction
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.75 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 23
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Dynamic Imaging Grade of Swallowing Toxicity
Description: The validated Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) will be performed on all collected videofluoroscopic swallowing studies to assess global swallowing function. The DIGEST total score is determined using the composite of individual airway safety and bolus efficiency subscores (range: 0-4). The DIGEST total is rated on a 5-point ordinal score ranging from 0 (no dysphagia) to 4 (life-threatening dysphagia).
Time Frame: Baseline; Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | ALS Individuals With Bulbar Dysfunction
Number analyzed (Participants) | 24
Participants
  Pre Nuedexta DIGEST 0 (Normal) | 3
  Post Nuedexta DIGEST 0 (Normal) | 7
Statistical Analysis 1: Comparison: ALS Individuals With Bulbar Dysfunction; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Speech Intelligibility
Description: The Sentence Intelligibility Test (SIT) will be performed to assess the change in speaking intelligibility over the 30 day period. The primary outcome of the SIT will be the percentage of sentence intelligibility (%) during oral reading.
Time Frame: Baseline; Day 30
Measure: Mean (Standard Error); unit: Percent Intelligibility
Arm/Group | ALS Individuals With Bulbar Dysfunction
Number analyzed (Participants) | 25
Percent Intelligibility
  Pre Nuedexta | 71.52 (6.62)
  Post Nuedexta | 73.06 (6.15)
Statistical Analysis 1: Comparison: ALS Individuals With Bulbar Dysfunction; Test type: Superiority; p = 0.647, Paired t test

3. Primary Outcome: Change in Patient-reported Outcome: Center for Neurologic Study-Bulbar Function Scale (CNS-BFS)
Description: The CNS-BFS is a validated patient-reported scale that assess self-reported impairments in the domains of speech, salivation and swallowing. Each domain contains 7 questions with ratings ranging from 1-5 with 5 considered the worst. For the speech domain, individuals who are unable to speak are assigned a value of 6 for each item (speech domain ranges from 1-6). Total scores ranging from 21 (no impairment) - 112 (severe impairment in all domains).
Time Frame: Baseline; Day 30
Measure: Mean (Standard Error); unit: Score
Arm/Group | ALS Individuals With Bulbar Dysfunction
Number analyzed (Participants) | 25
Score
  Pre Nuedexta | 56.87 (3.01)
  Post Nuedexta | 54.13 (2.97)
Statistical Analysis 1: Comparison: ALS Individuals With Bulbar Dysfunction; Test type: Superiority; p = 0.103, Paired t test

4. Primary Outcome: Change in ALSFRS-R Bulbar Subscale Score
Description: The ALS Functional Rating Scale-Revised Bulbar subscore is an outcome comprised of questions 1-3 on the validated ALSFRS-R scale. These items rate speech, swallowing and salivation functions on a scale from 0-total loss of function to 4- no symptoms for a total score of 0 to 12.
Time Frame: Baseline; Day 30
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ALS Individuals With Bulbar Dysfunction
Number analyzed (Participants) | 25
score on a scale
  Pre Nuedexta | 7.47 (0.38)
  Post Nuedextaa | 8.39 (0.37)
Statistical Analysis 1: Comparison: ALS Individuals With Bulbar Dysfunction; Test type: Superiority; p = 0.0004, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Bamboo Passage Reading Duration (in Seconds)
Description: The Bamboo Passage is a 60-word reading passage that is commonly used to measure speech duration.
Time Frame: Baseline; Day 30
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | ALS Individuals With Bulbar Dysfunction
Number analyzed (Participants) | 25
Seconds
  Pre Nuedexta | 66.19 (3.59)
  Post Nuedexta | 65.33 (3.59)
Statistical Analysis 1: Comparison: ALS Individuals With Bulbar Dysfunction; Test type: Superiority; p = 0.103, Paired t test

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of enrollment to study trial completion (30 days).
Arm/Group | ALS Individuals With Bulbar Dysfunction
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 4/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALS Individuals With Bulbar Dysfunction (N=28)
Prolonged hospitalization due to left leg DVT (General disorders) | 1 (1) — The subject was hospitalized for three days and treated for left leg DVT (unrelated to the study drug). The subject was treated accordingly and discharged home.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALS Individuals With Bulbar Dysfunction (N=28)
Fainting (General disorders) | 1 (1) — The subject reported a fainting episode, possibly related to the study drug. The subject discontinued participation in the study following this episode.
Diarrhea (Gastrointestinal disorders) | 1 (1) — The subject reported diarrhea for three days, possibly related to the study drug. The subject continued participating in the study.
Headache (General disorders) | 1 (1) — The study subject reported headaches over two days with a probable relationship to the study drug. The subject discontinued participation in the study.
Nausea (General disorders) | 1 (1) — The subject reported nausea for two days with a probable relationship to the study drug. The subject discontinued participation in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT03883581/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT03883581/ICF_001.pdf